CLINICAL TRIAL: NCT04350099
Title: Emotional Burden of Healthcare Professionals and the Epidemic Related to Covid Infection 19 -
Brief Title: Emotional Burden of Healthcare Professionals and Covid Infection 19
Acronym: Emocovid
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: 87RI20_0015/Emocovid
Record Dates: First submitted 2020-04-11; First posted 2020-04-16 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2020-04

CONDITIONS: Emotionnal Distress; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: quetionnary — Participants will complete self-questionnaires at different times during the epidemic

SUMMARY:
COVID-19 ( known as severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2)) has a highly polymorphic clinical presentation, ranging from pauci-symptomatic infection to severe, potentially complicated forms with acute respiratory distress syndrome or multisystemic organs failure. The picture may be initially severe, or it may progress in two stages, with worsening 7 to 10 days after the first symptoms with an overall case-fatality rate of 3 to 4%.

Its management is essentially symptomatic, as no antiviral treatment has so far demonstrated a clinical benefit in this condition.

In such a context, healthcare professionals assigned to COVID units will be faced with a heavy workload and emotional burden that could lead to psychological suffering or even burnout and its consequences.

We would therefore like to describe, using validated tools, the emotional evolution of the care workers at the Limoges University Hospital and the Esquirol University Hospital faced with this new pandemic infection. An initial and end-of-study evaluation of the caregivers will be carried out concerning their anxiety and depressive state, their personal capacity for resilience and their degree of empathy

ELIGIBILITY:
Inclusion Criteria:

* Health professional working in a COVID unit
* For the qualitative study: 24 participant selected at random to be interviewed

Exclusion Criteria:

* Refusal to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Health professional working
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-04-15 (Actual); Primary Completion 2021-02-15 (Estimated); Study Completion 2021-06-15 (Estimated)

PRIMARY OUTCOMES:
anxiety | 7 days,
  Assessing the anxiety of health professionals using Anxiety Disorder Assessment (GAD-7) scale.
  Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
anxiety | 15 days,
  Assessing the anxiety of health professionals using Anxiety Disorder Assessment (GAD-7) scale.
  Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
anxiety | 1 month
  Assessing the anxiety of health professionals using Anxiety Disorder Assessment (GAD-7) scale.
  Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
anxiety | 3 month
  Assessing the anxiety of health professionals using Anxiety Disorder Assessment (GAD-7) scale.
  Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CH Esquirol, Limoges
  - CHU de Limoges, Limoges
  - HCL LYON, Lyon